CLINICAL TRIAL: NCT01674582
Title: Treatment Effects Inclusive Cognitive Impact and Possibilities to Individually Adjusted Treatment in Patients With Intracranial Tumors With Clinical, Neuropsychological and Imaging Parameters.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version1.0
Record Dates: First submitted 2012-01-23; First posted 2012-08-29 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Intracranial Tumor
Keywords: Glioma; Brain tumors; Brain metastases; MRI; Cognitive measurement; Neuropsychological evaluation; DW-MRI; P-MRI; MRS
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI, Neuropsychological testing (Other)
  Interventions: Other: MRI, neuropsychological evaluation, blood sampling

INTERVENTIONS:
Other: MRI, neuropsychological evaluation, blood sampling — MRI at timepoints given above, neuropsychological testing after surgery, but before radiotherapy or chemotherapy.
  Neuropsychological testing month 3 during treatment. Neuropsychological testing after 1 year. Neuropsychological testing after 2 years.

SUMMARY:
The main purposes with this trial is to investigate the potential of MRI with diffusion and blood volume, flow in brain to diagnose and to measure treatment effects in patients with intracranial tumors, especially gliomas and metastases in a prospective trial, to evaluate the possibilities to individually adjusted treatment in this category of patients depending on treatment outcomes measured by MRI, to perform clinical follow up in connection with MRI to evaluate a correlation and to perform testing of cognitive ability before, during, and after treatment and to investigate if given treatment causes any decrease in the patients habitual state.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Suspected primary brain tumor, verified glioblastoma or non surgically treated metastases from solid tumor
* Increasing MRI changes in patients with previous verified glioblastoma
* Be able to speak Swedish without difficulties (because of the neuropsychological investigations)
* Written informed concent

Exclusion Criteria:

* Unability to perform MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Early prediction of treatment response based on MRI parameters. | Three weeks compared to baseline.

SECONDARY OUTCOMES:
Neuropsychological function. | Month 3, 12, and 18 compared to baseline
  Neuropsychological testing to evaluate the correlation between MRI results and neuropsychological status in participating patients. This applies for 80 patients of 150 of the patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Maly Sundgren, MD. PhD, Principal Investigator — Skåne University Hospital Lund
Locations (1):
- Lund University Hospital, Lund, Sweden